CLINICAL TRIAL: NCT01706016
Title: Local Treatment by Thermic Destruction of Primitive Breast Cancer. Phase II: Feasibility and Effectiveness, Standardization of Procedures.
Brief Title: Local Treatment by Thermic Destruction of Primitive Breast Cancer
Acronym: LASERBREAST1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A00448-35; 2011/1773 (Other: Institut Gustave Roussy)
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with breast cancer smaller than 20mm (Experimental)
  Interventions: Procedure: Thermic destruction of tissue by Laser using the Novilase device

INTERVENTIONS:
Procedure: Thermic destruction of tissue by Laser using the Novilase device

SUMMARY:
Demonstrate the effectiveness of laser in the treatment of cancerous lesions by determinating with histological analysis of the specimen the percentage of tumor cells remaining in the area treated by the laser

ELIGIBILITY:
Inclusion Criteria:

* Noninflammatory unilateral and unifocal breast cancer
* Size </= 20mm (ultrasound measure)
* Histological confirmation of cancer by biopsy grade status hormone and HER2.
* Good delineation of the lesion on ultrasound.
* Minimum distance of 5 mm between the tumor and the skin between the tumor and muscle.
* Age between 18 and 80
* ECOG performance status 0 or 1

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2012-10-09 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

PRIMARY OUTCOMES:
Effectiveness of laser treatment | 28 days after initial diagnosis
  Destruction of the carcinoma will be assess by histological analysis of the specimen.
  If more than 10% of viables cancerous cells are remaining in the volume treated by laser, the procedure would be a fail

SECONDARY OUTCOMES:
Life quality | D-0 and before the surgery
  Life quality will be assess using the questionnaire QLQ-C30 breast module BR23-version 3

CONTACTS AND LOCATIONS:
Overall Officials: Jean Remy GARBAY, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (3):
- France (3):
  - Centre Oscar Lambret, Lille, Nord
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - Hopital Lariboisière, Paris